CLINICAL TRIAL: NCT07365358
Title: A Multi-center, Randomized, Open-label, Active Comparator-controlled, Phase 4 Clinical Trial to Evaluate the Efficacy and Safety of Empagliflozin or Glimepiride Combination Therapy in Type 2 Diabetes Mellitus Patients Inadequately Controlled With Metformin and Sitagliptin
Brief Title: Evaluate the Efficacy and Safety of Empagliflozin or Glimepiride Combination Therapy in Type 2 Diabetes Mellitus Patients
Acronym: EMPAGO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B91_02DM2502
Record Dates: First submitted 2026-01-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Diabete Type 2
Keywords: Diabete Type 2; Empagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expermental group 1 (Experimental): Empamax® 10mg
  Interventions: Drug: empagliflozin 10mg
- Expermental group 2 (Active Comparator): Amaryl® 1mg
  Interventions: Drug: Glimepiride 1mg

INTERVENTIONS:
Drug: empagliflozin 10mg — once a day for 24 weeks
  Other Names: Empamax 10mg
  Arms: Expermental group 1
Drug: Glimepiride 1mg — once a day for 24 weeks
  Other Names: Amaryl 1mg
  Arms: Expermental group 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Empagliflozin or Glimepiride Combination Therapy in Type 2 Diabetes Mellitus Patients

DETAILED DESCRIPTION:
This study is a Multi-center, Randomized, Open-label, Active comparator-controlled, Phase 4 Clinical Trial to evaluate the efficacy and safety of Empagliflozin or Glimepiride Combination Therapy in Type 2 Diabetes Mellitus Patients

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years old
* Type 2 diabetes mellitus
* Patient who has been taking oral hypoglycemic agents for over 8 weeks
* Agreement with written informed consent

Exclusion Criteria:

* Type 1 diabetes mellitus or secondary diabetes mellitus
* Patients with complications of severe diabetes such as proliferative diabetic retinopathy
* Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Patients with abnormal laboratory test results according to the protocol
* Continuous or non-continuous treatment with insulin for over 7 days within 12 weeks prior to screening
* History of treatment with corticosteroids within 4 weeks prior to screening

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who meet 3 conditions at the same time | Baseline and Week 24
  1. No hypoglycemic events(<70mg/dL) for 24 weeks
  2. No weight change at 24 week
  3. HbA1c <7.0% at 24 week

SECONDARY OUTCOMES:
Percentage of subjects who meet 3 conditions at the same time | Baseline and Week 12
  1. No hypoglycemic events(<70mg/dL) for 12 weeks
  2. No weight change at 12 week
  3. HbA1c <7.0% at 12 week
Change from baseline in HbA1c and FPG | Baseline and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: In-Kyung Jeong, MD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No